CLINICAL TRIAL: NCT02344316
Title: Melatonin for Migraine Prevention in Adolescents: A Pilot Remote Trial: "The BRAiN-M Study"
Brief Title: Bringing Relief to Adolescents Naturally Using Melatonin for Migraine
Acronym: BRAiN-M
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amy Gelfand (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Sponsor-Investigator, Amy Gelfand, Assistant Professor of Neurology, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14-14251
Record Dates: First submitted 2015-01-12; First posted 2015-01-22 (Estimated); Results first posted 2021-09-09 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-08

CONDITIONS: Migraine in Adolescents
MeSH Terms: interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Melatonin (Active Comparator): Group randomized to melatonin 3 mg orally nightly
  Interventions: Drug: Melatonin
- Placebo (Placebo Comparator): Group randomized to placebo orally nightly
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Melatonin — Taken at 9 PM or 1 hour before bedtime, whichever is earlier
  Other Names: Rugby melatonin
  Arms: Melatonin
Other: Placebo — Matching placebo taken at 9 PM or 1 hour before bedtime, whichever is earlier
  Arms: Placebo

SUMMARY:
Migraine in adolescents is common and effective and safe preventive treatments are needed. This is a pilot randomized controlled trial of melatonin versus placebo for migraine prevention in adolescents 12-17 years old.

DETAILED DESCRIPTION:
This is a pilot randomized controlled trial of melatonin vs. placebo for migraine prevention in adolescents 12-17 years old. The main goal of this pilot study is to estimate variance in the outcome measures to help with planning the future fully powered study. Participants will have an in person enrollment visit, followed by phone follow up visits and headache diary data collection via smart phone or internet.

ELIGIBILITY:
Inclusion Criteria:

1. Age 12-17 years and weight ≥40 kg, to allow consistent dosing for all participants of the melatonin dose that has been found to be effective in adults
2. Resides in California
3. Headache fulfills International Classification for Headache Disorders, Third Edition (beta version)33 criteria for episodic migraine (with or without aura) in adolescents
4. Has been experiencing episodic headaches for at least six months
5. Experiences between 6-14 days of migraine/migrainous headaches per month at baseline (cutoff for chronic migraine is ≥15 days/month)
6. Developmentally able to provide age-appropriate level of assent
7. Has a parent/guardian capable of giving written informed consent
8. Has daily access to a smartphone in order to be able to complete daily study procedures such as diary completion, and to receive text reminders
9. Subject and parent agree the adolescent will not use over-the-counter melatonin, or another migraine preventive medication, while participating in the study
10. Participant and at least one parent speak English

Exclusion Criteria:

1. Currently (or within the last 4 weeks) using any medication or device with migraine preventive properties: i.e. topiramate, amitriptyline, nortriptyline, propranolol, metoprolol, sodium valproate, gabapentin, flunarizine, methysergide, riboflavin, butterbur, coenzyme Q10, or the Cefaly TENS device. For onabotulinum toxin, they will have to have been off it for at least three months
2. Use of other sleep medication or sedating medication, such as benzodiazepines, trazodone, or melatonin receptor agonists
3. History of allergy or adverse event with previous use of exogenous melatonin
4. Previous ineffective trial of melatonin 3 mg nightly for migraine prevention, where the trial duration was at least three months in duration
5. Inability to swallow pills, if this inability persists after instruction on pill-swallowing techniques
6. History of epilepsy or seizure
7. Overuse of acute headache medications, wherein medication overuse is defined33 as ≥4 days per month of barbiturate containing compounds, ≥10 days per month of opioid containing compounds, or ≥10 days per month of triptans or ergot-containing compounds. Those using non-specific analgesics ≥15 days per month would also be excluded
8. Adolescent does not have the cognitive capacity to give verbal assent to participate, or the investigator thinks the adolescent does not have the cognitive capacity to complete the diary, even with parental assistance
9. For females: Pregnancy, lactating or planning to become pregnant during the study. For males: planning to father a child during the study
10. Abnormal neurologic examination findings
11. Serious medical illness of any kind; seriousness as judged by the investigator
12. The investigator does not think the participant can comply with study procedures, or does not think it is medically appropriate for the participant to be in the study

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2015-05; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy A Gelfand, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - UCLA Headache Research and Treatment Program, Los Angeles, California
  - UCSF Pediatric Brain Center, San Francisco, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Masruha MR, Lin J, de Souza Vieira DS, Minett TS, Cipolla-Neto J, Zukerman E, Vilanova LC, Peres MF. Urinary 6-sulphatoxymelatonin levels are depressed in chronic migraine and several comorbidities. Headache. 2010 Mar;50(3):413-9. doi: 10.1111/j.1526-4610.2009.01547.x. Epub 2009 Oct 8. PMID 19817880
- [Background] Masruha MR, de Souza Vieira DS, Minett TS, Cipolla-Neto J, Zukerman E, Vilanova LC, Peres MF. Low urinary 6-sulphatoxymelatonin concentrations in acute migraine. J Headache Pain. 2008 Aug;9(4):221-4. doi: 10.1007/s10194-008-0047-5. Epub 2008 Jul 2. PMID 18594760
- [Background] Peres MF, Masruha MR, Zukerman E, Moreira-Filho CA, Cavalheiro EA. Potential therapeutic use of melatonin in migraine and other headache disorders. Expert Opin Investig Drugs. 2006 Apr;15(4):367-75. doi: 10.1517/13543784.15.4.367. PMID 16548786
- [Background] Peres MF, Zukerman E, da Cunha Tanuri F, Moreira FR, Cipolla-Neto J. Melatonin, 3 mg, is effective for migraine prevention. Neurology. 2004 Aug 24;63(4):757. doi: 10.1212/01.wnl.0000134653.35587.24. No abstract available. PMID 15326268
- [Background] Peres MF, Sanchez del Rio M, Seabra ML, Tufik S, Abucham J, Cipolla-Neto J, Silberstein SD, Zukerman E. Hypothalamic involvement in chronic migraine. J Neurol Neurosurg Psychiatry. 2001 Dec;71(6):747-51. doi: 10.1136/jnnp.71.6.747. PMID 11723194
- [Background] Fallah R, Shoroki FF, Ferdosian F. Safety and efficacy of melatonin in pediatric migraine prophylaxis. Curr Drug Saf. 2015;10(2):132-5. doi: 10.2174/1574886309666140605114614. PMID 24909684

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There was a 28 day baseline run-in prior to randomization.
Period: Overall Study
Arm/Group | Melatonin | Placebo
Started | 13 | 13
Completed | 12 | 11
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Melatonin | Placebo | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13 | 13 | 26
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15 (1.2) | 14.1 (1.7) | 14.5 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Migraine/Migrainous Days Per 28 Day Period
Description: Number of Migraine/Migrainous Days Per 28 Day Period in melatonin group and placebo group as measured using an online/mobile device headache diary.
Time Frame: final 4 weeks of treatment
Measure: Mean (Standard Error); unit: days
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 12 | 11
days | 3.6 (0.9) | 4.9 (1.7)

2. Secondary Outcome: Number of Minutes to Sleep Onset
Description: Number of minutes to sleep onset as measured by a FitBit.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 13 | 13
minutes | 15.2 (10.7) | 17.2 (12)

3. Secondary Outcome: Number of Participants Recruited From Each Recruitment Strategy
Description: Each recruitment strategy will be analyzed for number of participants successfully enrolled.
Time Frame: During the enrollment period, approximately 1 year
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: All Participants
Arm/Group | All Participants
Number analyzed (Participants) | 31
Participants
  Clinic recruitment | 6
  Newspaper advertising | 3
  Social media advertising (eg, Facebook and Google+ | 11
  Electronic medical record letter invitation | 10
  Other | 1

4. Secondary Outcome: Medication Adherence as Measured by Number of Openings Per Participant
Description: eCAP tack caps will be used to measure medication adherence and the number of openings will be recorded per participant.
Time Frame: during the "At Home Active Study Period" or Weeks 5-16
Measure: Mean (Standard Deviation); unit: Mean Number of Openings
Groups:
- Melatonin: Group randomized to melatonin 3 mg orally nightly Melatonin: Taken at 9 PM or 1 hour before bedtime, whichever is earlier
- Placebo: Group randomized to placebo orally nightly Placebo: Matching placebo taken at 9 PM or 1 hour before bedtime, whichever is earlier
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 12 | 12
Mean Number of Openings | 39 (27) | 60 (28)

5. Secondary Outcome: Headache Diary Compliance Rate
Description: Number of participants that had ≥85% headache diary compliance during weeks 12-16 of the study.
Time Frame: Weeks 12-16 of the study
Measure: Count of Participants; unit: Participants
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 12 | 11
Participants | 11 | 10

ADVERSE EVENTS:
Arm/Group | Melatonin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 6/13 | 4/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Melatonin (N=13) | Placebo (N=13)
Daytime tiredness (General disorders) | 2 (2) | 0 (0) — Daytime tiredness
Unscheduled medical visit for migraine (General disorders) | 2 (2) | 0 (0)
Low iron on routine labs (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Episode of vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1)
Accident (General disorders) | 0 (0) | 3 (3) — 1 kicked in the ribs 1 kicked in the testicle 1 passenger in a motor vehicle accident

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No